CLINICAL TRIAL: NCT00684580
Title: Protocol For Collecting Data On Patients With Childhood Cancer
Status: Recruiting | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SJLTFU
Record Dates: First submitted 2008-05-22; First posted 2008-05-26 (Estimated); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Childhood Cancer
Keywords: St. Jude Alumni; St. Jude Life Participants
MeSH Terms: conditions — Neoplasms | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational Group: Data Collection
  Interventions: Other: Data Collection

INTERVENTIONS:
Other: Data Collection — Continuing review of outcomes and late toxicities

SUMMARY:
Progress in the development of curative therapy for pediatric malignancies has resulted in increasing numbers of long-term childhood cancer survivors. This protocol is a means to provide continuing review of outcome and late toxicity for all patients actively being treated and previously treated for childhood cancer at St. Jude Children's Research Hospital.

DETAILED DESCRIPTION:
Previously at St. Jude Children's Research Hospital, monitoring and reporting of late treatment sequelae developing in protocol participants have occurred at the discretion of individual investigators. A formal mechanism for coordinating long-term follow-up data collection of late cancer-related toxicity did not exist within the institution, nor did a central data repository to facilitate correlation of clinical and treatment factors predisposing to toxicity. Central coordination of late effects monitoring and reporting at St. Jude offers the potential benefit of facilitating timely communication about life-threatening or unanticipated late toxicity to investigators developing contemporary therapeutic studies and monitoring predisposed survivors who may benefit from preventive or corrective interventions.

This study centralizes the late effects monitoring and reporting of St. Jude therapeutic studies which have been completed under the auspices of one umbrella protocol. This protocol is not an independent research study, but rather a means to aggregate outcome and late effects reporting regarding all patients actively being treated and previously treated at St. Jude Children's Research Hospital for the diagnosis of childhood cancer. Data collected on the patient will include only those data obtained through clinical staff or Cancer Registry encounters that are documented in the medical record or provided by the patient or family on follow-up forms. All monitored patients will have information provided regarding status (alive/expired), relapse, subsequent malignancies, and death for any cause. Clinical outcomes, toxicity and late effects monitoring planned in the study on which the patient was originally enrolled will be collected by the principal investigators of that study. Subjects will then be followed in the After Completion of Therapy on an annual basis for 10 years from diagnosis (or 10 years from completion of salvage therapy for relapse) or until they are at least 18 years of age. They will undergo specific screening laboratory, diagnostic imaging studies, and subspecialty consultations as medically indicated by predisposing cancer treatment exposures. At the time of discharge from ACT clinic the subject will begin annual lifetime follow-up by the St. Jude Cancer Registry.

ELIGIBILITY:
Inclusion Criteria:

* All St Jude patients actively being followed or treated for childhood cancer

Exclusion Criteria:

* St. Jude consult only patients
* St. Jude patients permanently discharged from care and follow-up Permanently discharged patients include patients who have electively transferred their oncologic care to another institution, those who are noncompliant with recommended follow-up or those leaving the institution against medical advice.
* Patients referred to St. Jude for limited care on phase 1 protocol.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients actively being treated and previously treated at St. Jude Children's Research Hospital for childhood cancer.
Sampling Method: Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2000-06-08 (Actual); Primary Completion 2045-05 (Estimated); Study Completion 2045-05 (Estimated)

PRIMARY OUTCOMES:
To provide continuing review of outcome and late toxicity for all patients actively being followed or treated for childhood cancer at St. Jude Children's Research Hospital, all St Jude Alumni and all St. Life participants. | 25 years

CONTACTS AND LOCATIONS:
Overall Officials: Melissa M Hudson, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols